CLINICAL TRIAL: NCT07352007
Title: A Prospective, Randomized Controlled, Phase II Study of Sintilimab Combined With Stereotactic Body Radiotherapy as Neoadjuvant Therapy for Resectable Hepatocellular Carcinoma
Brief Title: Sintilimab Combined With Stereotactic Body Radiotherapy as Neoadjuvant Therapy for Resectable Hepatocellular
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Lei ZHAO (Other)
Responsible Party: Sponsor-Investigator, Lei ZHAO, Shandong Cancer Hospital and Institute, Shandong Cancer Hospital and Institute
Organization: Shandong Cancer Hospital and Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Notable-HCC-II
Record Dates: First submitted 2026-01-11; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: HCC
MeSH Terms: interventions — sintilimab; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sintilimab +Stereotactic Body Radiotherapy +surgery (Experimental): Sintilimab 200 mg via intravenous infusion on day 1 of each 3-week cycle, for a total of two cycles. This will be combined with SBRT, administered as 8 Gy per fraction for 3 fractions on days 1, 3, and 5. Surgery will be performed 4-6 weeks after the last treatment, following the assessment of the patient's condition.
  Interventions: Procedure: SBRT; Drug: Sintilimab; Procedure: Surgery
- control (Other): Surgery
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: SBRT — SBRT :8 Gy per fraction for 3 fractions on days 1, 3, and 5.
  Arms: Sintilimab +Stereotactic Body Radiotherapy +surgery
Drug: Sintilimab — 200mg ivgtt,D1,Q3W
  Arms: Sintilimab +Stereotactic Body Radiotherapy +surgery
Procedure: Surgery — Surgery

SUMMARY:
This study is a prospective, randomized controlled, phase II trial evaluating the efficacy and safety of neoadjuvant therapy with Sintilimab combined with SBRT in patients with resectable hepatocellular carcinoma.

After meeting the inclusion and exclusion criteria and providing informed consent, eligible subjects will be randomly assigned to the experimental group or the control group:

* Experimental Group: Subjects will receive Sintilimab 200 mg via intravenous infusion on day 1 of each 3-week cycle, for a total of two cycles. This will be combined with SBRT, administered as 8 Gy per fraction for 3 fractions on days 1, 3, and 5. Surgery will be performed 4-6 weeks after the last treatment, following the assessment of the patient's condition. Postoperative adjuvant therapy with Sintilimab monotherapy (200 mg Q3W) will be administered until disease recurrence, death, intolerable toxicity, withdrawal of informed consent, initiation of new antitumor therapy, or other protocol-specified reasons occur, for a maximum of one year.
* Control Group:Subjects will undergo surgery directly. Postoperative adjuvant therapy with Sintilimab monotherapy (200 mg Q3W) will be administered until disease recurrence, death, intolerable toxicity, withdrawal of informed consent, initiation of new antitumor therapy, or other protocol-specified reasons occur, for a maximum of one year.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be provided and signed prior to the implementation of any trial-related procedures.
2. Male or female subjects aged ≥18 years and ≤75 years.
3. ECOG PS score of 0-1.
4. BCLC 0-B.
5. Diagnosed with HCC according to the diagnostic criteria of the Chinese Guidelines for the Diagnosis and Treatment of Primary Liver Cancer (2019 Edition).
6. CNLC Stage IA-IIB.
7. Child-Pugh score of ≤7.
8. No prior systemic antitumor therapy for hepatocellular carcinoma.
9. Assessed as suitable for R0 resection surgery.
10. Assessed as having no contraindications to SBRT and immunotherapy.
11. Estimated life expectancy of >3 months.
12. At least one measurable lesion according to RECIST 1.1 or mRECIST criteria.
13. Adequate organ and bone marrow function, defined as follows:a) Hematology: Absolute neutrophil count (ANC) ≥1.5×10⁹/L; Platelet count (PLT) ≥75×10⁹/L; Hemoglobin (HGB) ≥9.0 g/dL.b) Liver function: Serum total bilirubin (TBIL) ≤3 × upper limit of normal (ULN); Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase (ALP) ≤5 × ULN; Serum albumin ≥28 g/L.c) Renal function: Serum creatinine (Cr) ≤ 1.5 × ULN or creatinine clearance (CCr) ≥ 50 mL/min (Cockcroft-Gault formula); Urinalysis shows urine protein <2+; For patients with baseline urinalysis showing urine protein ≥2+, a 24-hour urine collection must demonstrate 24-hour urine protein <1 g.d) Coagulation function: International normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN.
14. For subjects with acute or chronic active hepatitis B or C infection, continuous antiviral therapy must be administered during the study period.
15. For female subjects of childbearing potential, a negative urine or serum pregnancy test must be confirmed within 3 days prior to receiving the first dose of the study drug (Cycle 1, Day 1). If a urine pregnancy test is inconclusive, a blood pregnancy test is required. Non-childbearing potential is defined as being post-menopausal for at least 1 year, or having undergone surgical sterilization or hysterectomy.
16. If there is a risk of conception, all subjects (both male and female) must use highly effective contraceptive methods (with a failure rate of <1% per year) throughout the entire treatment period and for at least 120 days after the last dose of the study drug (or 180 days after the last dose of chemotherapy). Estimated life expectancy ≥12 weeks.

Exclusion Criteria:

1. History of any histologically/cytologically confirmed malignancy other than HCC.
2. History of hepatic encephalopathy, or history of liver transplantation.
3. Presence of any extrahepatic metastatic lesions.
4. Prior receipt of any systemic antitumor therapy for HCC, including treatment with antibodies such as anti-PD-1, anti-PD-L1, or anti-CTLA-4 agents.
5. Acute or chronic active hepatitis B or C infection, defined as: Hepatitis B virus (HBV) DNA >2000 IU/mL or 10⁴ copies/mL; Hepatitis C virus (HCV) RNA >10³ copies/mL; Co-positive for Hepatitis B surface antigen (HBsAg) and anti-HCV antibody.
6. Radiotherapy received within 3 weeks prior to the first dose.
7. Human Immunodeficiency Virus (HIV) infection (positive HIV 1/2 antibodies) or known active syphilis infection.
8. Severe infections that are either active or poorly controlled clinically.
9. Active autoimmune disease that required systemic treatment within the past 2 years prior to the first dose.
10. Known history of primary immunodeficiency. The presence of autoimmune antibodies alone requires the investigator's judgment to confirm the presence of an autoimmune disease.
11. Use of immunosuppressive medication within 4 weeks prior to the first dose, with the exception of intranasal, inhaled, or other routes of locally administered corticosteroids, or systemic corticosteroids at physiological doses (i.e., not exceeding 10 mg/day prednisone or an equivalent dose of other corticosteroids). Temporary use of corticosteroids for conditions such as asthma or COPD for dyspnea is permitted.
12. Administration of any live attenuated vaccine within 4 weeks prior to the first dose or planned administration during the study period.
13. Any local therapy for liver cancer received within 4 weeks prior to the first dose.
14. Diagnosis of another malignancy within 5 years prior to the first dose, with the exception of radically treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and/or carcinoma in situ that has undergone radical resection. If another malignancy or HCC was diagnosed more than 5 years prior to the first dose, pathological or cytological confirmation is required for any recurrent or metastatic lesions.
15. Known allergy to any component of the Sintilimab formulation; or history of severe allergic reactions to other monoclonal antibodies or tyrosine kinase inhibitors.
16. Treatment received as part of another clinical trial within 4 weeks prior to the first dose.
17. Female patients who are pregnant or breastfeeding.
18. Any other acute or chronic disease, psychiatric disorder, or abnormal laboratory test value that may lead to the following outcomes: increased risk associated with study participation or study drug administration, interference with the interpretation of study results, and based on the investigator's judgment, makes the patient unsuitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-12-28 (Estimated); Primary Completion 2028-01-20 (Estimated); Study Completion 2031-01-20 (Estimated)

PRIMARY OUTCOMES:
Three-year recurrence rate | From date of resection until the date of first documented progression, assessed up to 3 years
  the proportion of individuals who experience their first radiological recurrence or death (whichever occurs first) from the time of enrollment in the group until the 3-year time point.

SECONDARY OUTCOMES:
Five-year recurrence rate | From date of resection until the date of first documented progression, assessed up to 5 years
  the proportion of individuals who experience their first radiological recurrence or death (whichever occurs first) from the time of enrollment in the group until the 5-year time point.
Recurrence free survival | From date of resection until the date of first documented progression, assessed up to 3 years
  the time from the end of treatment to tumor recurrence or patient death.
Overall survival (OS) | From date of resection until the date of death from any cause, assessed up to 5 years
  as the time from enrollment to the death of the subject for any reason
Pathologic complete response (pCR) | Up to one year
  The proportion of subjects whose postoperative pathological examination did not detect residual cancer cells

CONTACTS AND LOCATIONS:
Locations (1):
- ShandongShandong Cancer Hospital and Institute, Jinan, Shandong, China